CLINICAL TRIAL: NCT05854069
Title: Adapting FAMS to Optimize CGM Use Among Emerging Adults With Type 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); University of Utah (Other); University of California, Merced (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Lindsay Mayberry, Principle Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 220847; G-2203-05822 (Other Grant/Funding Number: The Leona M. and Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2023-04-24; First posted 2023-05-11 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
Keywords: Continuous glucose monitor; Social support; Goal setting; Diabetes distress; Hemoglobin A1c; Time in range; Emerging adults; Family support; Text message; Mobile health
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAMS-T1D (Experimental): Participants will receive FAMS-T1D components (monthly phone coaching and text message support for goals) for 6 months. Support persons will receive text messages that are tailored to the goal set by the person with type 1 diabetes.
  All persons with diabetes will receive text messages regarding how to access their HbA1c results and receive links providing information to assist them in self-care behaviors related to their diabetes. All support persons will also receive materials about type 1 diabetes and how to provide helpful support to the person with diabetes.
  Interventions: Behavioral: FAMS-T1D; Behavioral: Digital resources for diabetes
- Digital resources for diabetes (Placebo Comparator): All persons with diabetes will receive text messages regarding how to access their HbA1c results and receive links providing information to assist them in self-care behaviors related to their diabetes. All support persons will also receive materials about type 1 diabetes and how to provide helpful support to the person with diabetes.
  Interventions: Behavioral: Digital resources for diabetes

INTERVENTIONS:
Behavioral: FAMS-T1D — FAMS-T1D involves monthly phone coaching that assists individuals in setting specific and time bound diabetes goals with automated text message support to the patient participant and less frequent automated text messages to their support person, if one is enrolled.
  Behavioral: Diabetes Resources High quality digital materials about diabetes management will be provided upon enrollment and send to participants quarterly.
  Other Names: Family/friend Activation to Motivate Self-Care for those with Type 1 Diabetes
  Arms: FAMS-T1D
Behavioral: Digital resources for diabetes — Quality digital resources about diabetes management provided upon enrollment and during the study.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of an adapted FAMS (Family/friend Activation to Motivate Self-care) intervention on CGM use among study participants who are CGM users. We will leverage the infrastructure of an NIDDK-funded RCT evaluating FAMS-T1D among N=280 emerging adults with T1D who have elevated hemoglobin A1c or elevated diabetes distress (NCT05820477). We anticipate at least 50% using CGM to be included in these analyses.

DETAILED DESCRIPTION:
FAMS (Family/friend Activation to Motivate Self-care) is a mobile phone-delivered intervention, based on Family Systems Theory, which helps adults with diabetes set behavioral goals and improve support received from friends and family for goal success. FAMS includes monthly phone coaching and text message support by FAMS coaches for the person with diabetes (PWD) and the option to enroll a support person (SP) to receive automated texts tailored to the self-care goals the person with T1D sets in coaching sessions. Adaptations specific to CGM include the option to set CGM use goals in coaching (and receive associated text support) and skill-building exercises during coaching to support data sharing relationships (e.g., establishing, setting and adjusting ground rules about communication).

Within the FAMS-T1D RCT (NCT05820477), we will test effects of FAMS-T1D on CGM use use relative to enhanced treatment as usual. We will evaluate effects on CGM use from baseline to post-intervention (6 months) as the primary endpoint. Study start date for the nested trial (NCT05854069) is the enrollment date of the first participant using a CGM. Since the goal of this trial is to assess effects of the adapted FAMS intervention on CGM use, the date participant CGM usage was confirmed is considered the enrollment date.

ELIGIBILITY:
Inclusion Criteria:

PERSONS WITH DIABETES

* Ages 18-24
* Have a diagnosis of T1D and has been taking insulin for at least one year
* Comfortable sending and receiving texts
* Can speak, read, and write in English
* Meets one of the following two criteria: 1) has a most recent A1c value in the EHR that is 7.5% or higher (or missing) OR 2) screen positive for diabetes distress on the two-item Diabetes Distress Screen (DDS-2)
* Using a continuous glucose monitor (CGM)

SUPPORT PERSONS

* Age 18 or older
* Can speak, read, and write in English or Spanish
* Comfortable sending and receiving texts

Exclusion Criteria:

PERSONS WITH DIABETES

* Has a condition that would prohibit study completion (intellectual disability, blindness or auditory limitations, severe mental illness)
* Plans to live outside the country during the study period

SUPPORT PERSONS

* Shares a phone with the person with diabetes
* Plans to live outside of the country during the study period

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
CGM frequency of use during the intervention period | Baseline and 6 months post-baseline
  Change in CGM frequency of use assessed by self-report on questionnaire; more frequent use/higher is better
CGM frequency of use during the intervention period | Baseline and 6 months post-baseline
  Change in CGM frequency of use assessed by objective CGM data (% of time; higher is better)
Gaps in CGM use | 6 months post-baseline
  Length of gaps in CGM use as assessed by objective CGM data (measured in number of consecutive days without CGM data; higher is worse)

SECONDARY OUTCOMES:
CGM behavioral responses during the intervention period | Baseline and 6 months post-baseline
  Change in frequency of making behavioral changes in response to CGM data assessed by self-report; higher scores indicate more frequent response (better)
Barriers to CGM use during the intervention period | Baseline and 6 months post-baseline
  Change in perceived influence of CGM on glycemic control scale assessed by Glucose Monitoring Survey; higher scores indicate more perceived problems with CGM use (worse)
Barriers to CGM use during the intervention period | Baseline and 6 months post-baseline
  Change in perceived influence of CGM on social complications assessed by Glucose Monitoring Survey; higher scores indicate more perceived problems with CGM use (worse)
CGM satisfaction during the intervention period | Baseline and 6 months post-baseline
  Change in CGM satisfaction assessed by Benefits of CGM scale; higher scores indicate more perceived benefits of CGM use (better)

OTHER OUTCOMES:
Data sharing during the intervention period | 6 months post-baseline
  Number of data sharing relationships, between groups; more is better
Satisfaction with data-sharing relationships | 6 months post-baseline
  Satisfaction with data-sharing relationships assessed by CGM-Satisfaction Scale; higher scores are better

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published, de-identified data will be available upon requests made to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study results are posted on clinical trials and outcomes published in a peer-reviewed journal, until 5 years later.
Access Criteria: Contact the principal investigator